CLINICAL TRIAL: NCT02438527
Title: Flowchart-Assisted Resuscitation. Standard CPR vs. Chest Compressions Only: What Happened to the Quality?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Bernhard Roessler, PD Dr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 20151136
Record Dates: First submitted 2015-04-29; First posted 2015-05-08 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: CPR Guidelines

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chest Compressions Only (Experimental): After recruitment and consenting, volunteers in the "chest compressions only" arm will receive a chart with a description of Basic Life Support without mouth to mouth ventilations. The participants will be asked to perform Cardiopulmonary Resuscitation according to the chart for a period of 5minutes on a manikin in a simulated cardiac arrest scenario.
  Interventions: Behavioral: Chart for CPR guidance
- Standard CPR (Experimental): After recruitment and consenting, volunteers in the "standard CPR" arm will receive a chart with a description of Basic Life Support. The participants will be asked to perform Cardiopulmonary Resuscitation according to the chart (including the initial check, chest compressions and mouth to mouth ventilations) for a period of 5minutes on a manikin in a simulated cardiac arrest scenario.
  Interventions: Behavioral: Chart for CPR guidance

INTERVENTIONS:
Behavioral: Chart for CPR guidance

SUMMARY:
ABSTRACT

Background:

More than two thirds of sudden cardiac arrests are witnessed by bystanders. Bystander cardiopulmonary resuscitation (CPR) doubles survival from cardiac arrest. Importantly, even in witnessed cardiac arrests only 20% of the bystanders commence basic life support. Common reasons for not commencing include panicking and the perceived inability to perform CPR correctly. A meta-analysis could demonstrate that a simplification of the algorithm (compression-only dispatcher-assisted bystander CPR) led to a 22% increase in survival-to-hospital discharge. A recently published trial of the research group could demonstrate that the presence of a flowchart has a positive effect on the quality of BLS while at the same time increasing the rescuers' confidence. Nonetheless, performing CPR is exhausting. Previous publications have emphasized increasing fatigue with the duration of CPR efforts in both, standard and chest compressions-only CPR. Consequently, we wanted to test the hypothesis that chest compressions (CC) are delivered more correctly regarding the depth when utilizing the standard BLS algorithm with the aid of a flowchart as compared to the CC only algorithm utilizing an adapted CPR flowchart in a manikin resuscitation model.

Methods:

After consent of the Research Ethics Board of Medical University of Vienna and obtaining written informed consent of the participants, 84 medically untrained laypersons will be randomised to perform flow-chart assisted CPR for 300s following standard CPR guidelines or CC only CPR. The primary outcome parameter will be the total number of CC achieving the correct depth of 50-60mm. Secondary outcome parameters will be hands-off time, the total number of CC, and the compression rate. The total number of delivered rescue breaths, tidal volume, and time to deliver these will also be evaluated. Furthermore, the subjective point of exhaustion affecting the CPR quality, the reason for discontinuation of CPR if stopped within the 300sec. period and the exhaustion at the end of the CPR measures will be evaluated.

DETAILED DESCRIPTION:
Study Design The investigation will be conducted as a prospective, randomized controlled study performed by the Department of Anaesthesia, General Intensive Care and Pain Management, Medical University of Vienna, Austria, according to the Good Scientific Practise guidelines of the Medical University of Vienna. The data collection will be conducted in cooperation with the Training Centre of St. John Ambulance, Vienna, Austria.

Study Population Eligible are all volunteers of ≥18 years of age of non-medical profession, irrespective of gender. Exclusion criteria are professional medical training (nurses, medical doctors, physiotherapists, ergotherepeuts, emergency medical technician or equivalent), pregnancy (as by verbal response at the time of recruitment), and parallel participation in a clinical trial, or physical impairment or illness prohibiting physical effort.

Withdrawal and replacement of subjects

Subjects must be withdrawn under the following circumstances:

* at their own request
* if the subject violates the conditions laid out in the consent form/information sheet or disregards instructions by the study personnel

In all cases, the reasons why subjects are withdrawn must be recorded in detail in the case report form. Should the study be discontinued prematurely, all study materials (completed, partially completed and empty case report forms) will be retained.

Subjects who do not complete the study according to protocol will be replaced. The data from the replaced subjects will be eligible for analysis of the conducted trial periods and for safety variables.

Methodology

Sample Size In order to detect a clinically important difference of 20% in compression depth with a power of 0.8 and a significance level set at 0.05, the sample size calculation yielded a total needed number of participants at 74. Since a drop out rate of approx. 10% must be expected 84 participants will be recruited. Data regarding compression depth utilizing standard CPR techniques in a manikin model (43±12mm) were provided by a previous publication and used to estimate the sample size [Rössler et al. 2013]

Statistical Methods

Outcome parameters:

The primary outcome is total number of CC achieving the correct depth of 50-60mm in five minutes of manikin CPR. With this the authors want to test the hypothesis that chest compressions are delivered more correctly regarding the depth when utilizing the standard BLS algorithm with the aid of a flowchart as compared to the CC only algorithm utilizing an adapted BLS flowchart in a manikin resuscitation model. The secondary outcome parameter is hands-off time (HOT), which is defined as the sum of total time elapsed during the 300sec. of BLS in which no chest compressions are provided. This includes the pre-compression interval where the initial steps of BLS are performed as well as all interruptions of the CC, e.g. in order to ventilate or pause due to any other reason including exhaustion. Furthermore, the total number of CC, and the compression rate will be evaluated. The total number of delivered rescue breaths, tidal volume, and time to deliver these will also be evaluated.

Furthermore, questions regarding following points will be raised: "During CPR and without stopping your actions, please tell us "NOW" when you perceive your fatigue is affecting the quality of the life support performed", "How exhausted are you now (question raised directly after discontinuing the CPR) [McDonald et al. 2013] (Lickert Like Scale 1-10). If a participant choses to abort resuscitation attempts the open ended question "Why did you discontinue the resuscitation attempts?" will be raised.

Data management and calculations Data will be described as absolute frequencies and percentages for categorical data and using mean and standard deviations (SD) for normally distributed data. All tests for p-values are two-sided and p≤0.05 will be regarded to be statistically significant. Students t-test and chi-sqare test will be used as appropriate. As it is common practice, results of Likert-like scales will be treated as interval-measures and thereby analysed by using parametric tests [Norman et al. 2010, Cariio et al. 2008]. Local data management will be done using Microsoft Excel for Mac (Microsoft Corporation, USA) and R for Mac (R Foundation for Statistical Computing, Vienna, Austria) for statistical analysis. [R_Development_Core_Team 2009] Graphics will be created using PraphPad Prism for Mac (GraphPad Software Inc., La Jolla, USA).

Description of study days Volunteers will be invited to participate in the trial by the study personnel. Recruitment will be conducted at a Training Centre of St. John ambulance, Vienna, Austria, before the starts of the lessons. After giving written informed consent, participants will be randomized using a web based randomization program (www.random.org) and allocated to perform standard CPR or CC only. The randomization for group allocation will be kept in opaque and sealed envelopes.

The evaluation will be performed with an independent investigator using a computer attached Resusci-Anne Skillreporter by Laerdal-Medical® and the Laerdal Skillreporter Software with Segstat (Version 2.3.0, Laerdal Medical, Stavanger, Norway).

The participants will be asked to perform BLS for five minutes on a manikin. The participants will then be asked to undertake any action they deem necessary to rescue the person simulated by the resuscitation manikin. Participants will not be informed about the underlying hypothesis or the outcome parameters. The room will be prepared to minimise outside interruptions.

Additionally, participants will be instructed to indicate the point in time during CPR when they feel that their fatigue is affecting the quality of the life support performed. ("During CPR and without stopping your actions, please tell us "NOW" when you perceive your fatigue is affecting the quality of the life support performed.)

Participants in both groups will receive one of the charts right at the beginning of the scenario with the information that "this chart will provide information on how to perform CPR" and with the start of the clock further instructions regarding is content. Both groups will not receive any further introduction or support. At the beginning of the scenario, the manikin will be positioned in a supine position on the floor. There will be no clock visible for the participant while performing CPR. An investigator is acting as bystander able to call the emergency medical service or to be sent to look for an automated external defibrillator (which will not be available in the scenario). Nonetheless, the investigator is instructed not to provide any information on how to perform CPR and does not physically take part in the primary check, CC, or mouth-to-mouth ventilations.

Data of steps performed or left out will be documented in hardcopy on the case report form by an investigator and the exact times and details of chest compressions and ventilations will be documented electronically (Laerdal Skillreporter Software with Segstat (Version 2.3.0, Laerdal Medical, Stavanger, Norway)). Checklists of necessary steps will be created based on the ERC BLS Guidelines 2010 in the same manner as published previously [Roessler et al. 2007, Koster et al. 2010].

After the five-minute period has ended, the participants will be informed that the emergency medical service is now taking over and that they can stop performing CPR. Directly thereafter, they will be asked the following questions "How exhausted are you now on a scale from 1 to 10, where 1 indicates no exhaustion at all and 10 maximum exhaustion?" (Lickert Like 1-10). If a participant choses to abort resuscitation attempts before the five minutes are over, the open-ended question "Why did you discontinue the resuscitation attempts?" will be raised.

Risk/benefit assessment:

Apart from physical strain such as muscle pain or abrasion on the palm of the hand or knee after delivering chest compressions, there is no direct risk as the consequence of participation in the trial. To ensure participants added value, detailed information about the ERC CPR algorithm will be given after data collection. This information included written material on the 2010 CPR guidelines, or the 2015 CPR guidelines when available.

ELIGIBILITY:
Inclusion Criteria:

≥18 years of age

Exclusion Criteria:

* professional medical training (nurses, medical doctors, physiotherapists, ergotherepeuts, emergency medical technician or equivalent)
* pregnancy (as by verbal response at the time of recruitment)
* parallel participation in a clinical trial
* physical impairment or illness prohibiting physical effort.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2015-05-15 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
total number of CC achieving the correct depth of 50-60mm. | 5min. CPR

SECONDARY OUTCOMES:
hands-off time | 5min CPR
the total number of CC | 5min CPR
compression rate | 5min CPR